CLINICAL TRIAL: NCT01164267
Title: A Multicenter Phase II Study to Evaluate the Clinical Activity and the Safety Profile of Everolimus (RAD001) in Marginal Zone B-cell Lymphomas (MZL) EudraCT Number 2009-011725-14
Brief Title: Multicenter Phase II Study to Evaluate the Clinical Activity and the Safety Profile of Everolimus in Marginal Zone B-cell Lymphomas (MZL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IELSG 34; 2009-011725-14 (EudraCT Number)
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2012-05

CONDITIONS: Marginal Zone B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Everolimus — Everolimus (tablets, 5 mg) is given orally at the dose of 10 mg/day from day 1 to day 28 of each cycle for up to a total of 6 cycles or until progression. Patients with CR or PR may continue treatment until PD if well tolerated

SUMMARY:
This is a multicenter open-label uncontrolled phase II study. There are no previous clinical data to estimate the expected response rate of everolimus in MALT lymphomas and in the other less common MZLs (i.e. nodal and splenic) refractory or relapsing after at least 1 prior systemic treatment (chemotherapy or immunotherapy).

The primary objective of this study is to define the antitumor activity, in term of overall response rate (ORR), as sum of complete remissions (CR) and partial remissions (PR) of everolimus in relapsed or refractory marginal zone B-cell lymphomas.

The secondary objectives of this study are to assess safety, as acute or long-term toxicity, response duration (RD) (time to relapse or progression) in responders and progression-free survival (PFS) (time to disease progression or death from any cause) in all patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven diagnosis of marginal zone B-cell lymphoma relapsing/refractory following at least 1 prior systemic treatment (chemotherapy and or monoclonal antibodies).
2. Any stage (Ann Arbor I-IV).
3. No evidence of histologic transformation to aggressive lymphoma.
4. Measurable or evaluable disease.
5. Age > 18 years.
6. Life expectancy of at least 3 months.
7. ECOG performance status 0-1.
8. No prior diagnosis of neoplasm within 5 years, except cervical type 1 intraepithelial neoplasia or localized non-melanomatous skin cancer.
9. In case of prior diagnosis of solid organ tumors, no treatment over the last 5 years ond no current evidence of disease.
10. No prior chemo-or radiotherapy in the last 6 weeks, no prior immunotherapy in the last 8 weeks, no corticosteroids during the last 4 weeks unless low-dose prednisone chronically administered for indications other than lymphoma or lymphoma-related symptoms.
11. No major impairment of bone marrow function, renal function or liver function unless due to lymphoma.
12. No evidence of active opportunistic infections, no HIV infection, no evidence of HBV infection, no active HCV infection.
13. Women of childbearing potential are using effective contraception, are not breast feeding, are not pregnant and agree not to become pregnant during participation in the trial and during the 12 months thereafter. A negative pregnancy test is mandatory for all patients < 50 years (unless considered unnecessary by the investigator).

    Men agree not to father a child during participation in the trial and during the 12 months thereafter.
14. No serious cardiac, neurological or psychiatric disorders potentially hampering compliance with the study protocol and follow-up schedule.
15. Fasting serum cholesterol ≤ 200 mg/dL or ≤ 5 mmol/L AND fasting triglycerides ≤ 200 mg/dL. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
16. Written informed consent.

Exclusion Criteria:

1. Patients with newly diagnosed MZL.
2. Patients with concomitant or past hematological malignancies.
3. Presence or history of CNS lymphoma localization (either parenchymal or meningeal disease).
4. Cardiovascular disease (congestive heart failure; NYHA III or IV), unstable angina pectoris, significant cardiac arrhythmias requiring chronic treatment, or prior history of myocardial infarction in the last 3 months.
5. Serious underlying medical condition which could impair the ability of the patient to participate in the trial (e.g. uncontrolled diabetes mellitus, gastric ulcers, active autoimmune disease, ongoing infection e.g. HIV, hepatitis).
6. Concurrent anticancer drugs / treatments and experimental drugs. Previous radiation is allowed, unless the indicator lesion(s) are in the irradiated field.
7. Previous organ transplantation
8. Participation in another clinical trial within 30 days prior to trial entry
9. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Total Body CT-Scan | Every 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Zucca, MD, Study Chair — IOSI; Annarita Conconi, MD, Study Chair — AOU Maggiore della Carità Novara
Locations (10):
- General Hospital AKH, Vienna, Austria
- Italy (8):
  - Policlinico S. Orsola Malpighi, Bologna
  - Humanitas, Milan
  - San Raffaele Hospital, Milan
  - IEO, Milan
  - INT, Milan
  - AOU Maggiore della Carità, Novara
  - IRCCS Policlinico S. Matteo, Pavia
  - AOU S. Giovanni Battista, Torino
- IOSI, Bellinzona, Switzerland

REFERENCES:
- See also: Related Info — http://www.ielsg.org